CLINICAL TRIAL: NCT04007497
Title: Reconstruction of Hand and Upper Extremities Defects by Thin Random Pedicle Abdominal Flaps, Still a Valid Option in Developing Countries: A Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Saif Aldeen AlRyalat, Doctor in medicine, University of Jordan
Other Study IDs: UJordan plastic
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Upper Extremity Defects

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Traumatic defects of the soft tissues of the hand and upper extremities are common and may be challenging to the reconstructive surgeon. Several reconstructive procedures have been described to manage these defects, including local, regional, distant, and free flaps. The aim of this study is to report the techniques, outcomes, and complications of pedicle abdominal flaps in reconstructing hand and upper extremity defects. We included patients with different traumatic defects in the hand and upper extremities who underwent reconstruction by random pedicle abdominal flaps between 2002 and 2017. Data was collected and analyzed, variables studied included; patient age and sex, etiology and size of the defect, complications, outcomes, and the need for further revision procedures. Potential factors affecting flap survival were examined using appropriate statistical analysis.

DETAILED DESCRIPTION:
Traumatic soft tissue defects of the hand and upper extremity are common and may be challenging to the reconstructive surgeon, especially when they are severe and associated with exposed vital structures such as tendons, nerves, bones, and joints. Although these defects are rarely lethal; they are invariably resource demanding, and a source of significant long-term disability. Several reconstructive procedures have been described to cover hand and upper extremities soft tissue defects, including local, regional, distant, and free flaps. Traditionally, pedicle abdominal flaps, whether axial or randomly based, have been considered the standard for successful upper limb reconstruction.

With the introduction of microsurgery in the seventies of the last century, microsurgical free tissue transfers have become the gold standard for upper extremities functional reconstruction. Free flaps and other microsurgical techniques have been used to achieve early, functional, custom-tailored reconstructive solutions for upper limbs injuries. However, despite the superiority of free flaps, this option may not be always accessible especially in developing countries, owing to the high cost and technical demands. Moreover, they may be contraindicated in certain circumstances. In these situations, pedicle abdominal flaps may once again come into the light as an alternative option for safe and effective upper extremities reconstruction.

At Jordan University Hospital, with limited microsurgical facilities, the investigators have been using random pedicle abdominal flaps in patients with different traumatic hand and upper extremities defects. The aim of this retrospective study is to report the investigator's experience in using this technique, in regards to the indications, complications, outcomes, and evaluating factors affecting flap survival rate.

ELIGIBILITY:
Inclusion Criteria:

* different traumatic defects in the hand and upper extremities who underwent reconstruction by random pedicle abdominal flaps

Exclusion Criteria:

* Patients with incomplete data about the patient and the surgery

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with different traumatic defects in the hand and upper extremities who underwent reconstruction by random pedicle abdominal flaps.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
Reconstruction of hand and upper extremities defects by thin random pedicle abdominal flaps | 2002 and 2017
  The investigators will examine success rate of randome abdominal flap in managing upper extremity's defects

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, Amman, Jordan